CLINICAL TRIAL: NCT02620683
Title: Comparison of Buffered vs. Non-Buffered Lidocaine Used in Dental and Oral Surgical Procedures: Clinical Outcomes
Brief Title: Clinical Outcomes of Buffered vs. Non-Buffered Lidocaine
Acronym: BUFFL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Dental Foundation of North Carolina, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 15-1741; CHDEN 29920, D0117439000 (Other: Dental Foundation of North Carolina, Inc.)
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-10

CONDITIONS: Blood Levels of Buffered vs Non-buffered Lidocaine; Anesthetics, Local
Keywords: lidocaine, jaw
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buffered Lidocaine (Active Comparator): In week One each subject would receive anesthetic to block the inferior alveolar and lingual N; Halstead or Gow-Gates techniques. No Buccal N. block.
  Venous blood samples would be drawn from the antecubital fossa 30min post oral injection and assayed for blood lidocaine levels
  Interventions: Drug: Lidocaine
- Non-buffered Lidocaine (Active Comparator): In week One each subject would receive anesthetic to block the inferior alveolar and lingual N; Halstead or Gow-Gates techniques. No Buccal N. block. At least a week later injections would involve the alternate local anesthetic combination.
  Venous blood samples would be drawn from the antecubital fossa 30min post oral injection and assayed for blood lidocaine levels
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — See above
  Other Names: Xylocaine

SUMMARY:
Anecdotal reports suggest buffering lidocaine with epinephrine just before intraoral injection reduces time of onset, results in a deeper anesthetic effect, without the "sting" with injection from a low pH. Additional data are needed to establish clinical important outcomes such as the peak blood level of lidocaine as compared to the non-buffered drug combination.

Clinical pilot studies are proposed as the start of a series of investigations to support or modify the use of the buffered anesthetic for intraoral procedures.

DETAILED DESCRIPTION:
Specific Aims:

Compare blood levels at 30min post injection mandibular block with buffered and non- buffered 2% lidocaine with 1/100k epinephrine. Assess outcomes (pain levels during and post-injection, and onset of anesthesia symptoms) after buffered and non-buffered oral administration of 2% lidocaine with 1/100k epinephrine. Assess possible topical anesthetic properties of buffered and non-buffered oral administration of 2% lidocaine with 1/100k epinephrine

Hypotheses:

No difference in peak blood levels exist between buffered and non-buffered intraoral injection of 2% lidocaine with 1/100k epinephrine.

Injection of buffered local anesthetic will produce less discomfort for the subject as compared to the drug with a low pH.

Buffered local anesthetic will not produce a topical anesthetic effect

Study Time Frame: 6 months Month One IRB approvals. Recruit volunteers as subjects. Prepare case-books. Months Two-Three Clinical Study Months Four-Five Analyze Lab, QOL data Month Six Prepare Abstracts, Papers

Methods: Blinded, Randomized Clinical Design Recruit subjects with IRB approved consent at UNC Target enrollment 24 subjects Subjects will serve as their own controls in a cross-over AB/BA study design which is uniform within sequences, uniform within periods, and balanced Sample size justification: Primary interest is estimation of effect size from pilot study. 24 subjects should be sufficient to provide data to assess whether a larger study is warranted and provide estimates for sample size calculation for larger studies. Vital signs recorded: 10 min before, during at 30min intervals and after post-anesthetic clinical signs disappear: targeted lower lip no longer numb. Randomized subjects to be injected alternatively with 4cc of buffered and 4cc non-buffered oral administration of 2% lidocaine with 1/100k epinephrine.

SAS will be used to create randomization schedules:

The randomization will be performed first to type of drug given with a balanced randomization (half subjects buffered; half to non-buffered) An OMS resident, Dr Phero, will administer the drugs in the OMS clinic.

In week One each subject would receive anesthetic to block the inferior alveolar and lingual N; Halstead or Gow-Gates techniques. No Buccal N. block. At least a week later injections would involve the alternate local anesthetic combination.

Venous blood samples would be drawn from the antecubital fossa 30min post oral injection and assayed for blood lidocaine levels Timed Assessment: pre, during injection, and post-anesthetic for Clinical Onset of Anesthesia Signs: subject reported molar area numbness and numb lower lip on ipsilateral injected side. Assessment for pain level on injection; modified Likert-type scale

In addition at each clinic session an assessment of a topical anesthetic effect on contralateral lower lip with 5 drops of the injected drug placed on the clinically dry lower lip mucosa, Outcome yes/no.

Data Collection: UNC OMS clinic Venous blood samples (10cc) will be drawn from the antecubital fossa 30min post oral injection. Timed assessment pre, during injection, and post-anesthetic clinical Signs: molar area anesthesia, incisor area anesthesia, and numb lower lip for topical

Data Collection/Analysis:

Data will be managed by study staff. Data collection forms and questionnaires for clinical data will be developed to use Teleform for direct scanning input into an ACCESS database. Similar forms have been used in previous studies. All databases are stored on a password protected School of Dentistry server with specific group assignment. SAS will be used for database management and statistical analysis. Descriptive statistics are used to verify correct entry through range and logical checks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30 years
* ASA I
* Willingness to complete QOL instrument
* Willingness to participate in two sessions

Exclusion Criteria:

* Allergy to lidocaine class of anesthetic drugs
* Local anesthetic drug use in past week
* Current symptoms teeth or oral mucosa

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2015-12; Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond P White, Jr, DDS, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC School of Dentistry, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Phero JA, Nelson B, Davis B, Dunlop N, Phillips C, Reside G, Tikunov AP, White RP Jr. Buffered Versus Non-Buffered Lidocaine With Epinephrine for Mandibular Nerve Block: Clinical Outcomes. J Oral Maxillofac Surg. 2017 Apr;75(4):688-693. doi: 10.1016/j.joms.2016.09.055. Epub 2016 Oct 8. PMID 27815105

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Beginning in December 2015 23 subjects recruited for study conducted in the surgery clinic at UNC School of Dentistry
Pre-assignment Details: No enrolled subjects excluded.
Groups:
- Buffered Lidocaine, Then Non-buffered Lidocaine: At Visit 1 each subject received Buffered Lidocaine anesthetic to block the inferior alveolar and lingual N; using Halstead or Gow-Gates techniques. No Buccal N. block. Venous blood samples were drawn from the antecubital fossa 30min post oral injection and assayed for blood lidocaine levels. Following a 2-week washout, subjects received Non-buffered Lidocaine in the same fashion at Visit 2.
- Non-buffered Lidocaine, Then Buffererd Lidocaine: At Visit 1 each subject received Non-Buffered Lidocaine anesthetic to block the inferior alveolar and lingual N; using Halstead or Gow-Gates techniques. No Buccal N. block. Venous blood samples were drawn from the antecubital fossa 30min post oral injection and assayed for blood lidocaine levels. Following a 2-week washout, subjects received Buffered Lidocaine in the same fashion at Visit 2.
Period: First Intervention (Visit 1)
Arm/Group | Buffered Lidocaine, Then Non-buffered Lidocaine | Non-buffered Lidocaine, Then Buffererd Lidocaine
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0
Period: Washout (2 Weeks)
Arm/Group | Buffered Lidocaine, Then Non-buffered Lidocaine | Non-buffered Lidocaine, Then Buffererd Lidocaine
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0
Period: Second Intervention (Visit 2)
Arm/Group | Buffered Lidocaine, Then Non-buffered Lidocaine | Non-buffered Lidocaine, Then Buffererd Lidocaine
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Subjects who were randomized to receive either Buffered or Non-Buffered Lidocaine
Arm/Group | All Study Participants
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 21 [20 to 22]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Lidocaine Blood Levels 30 Minutes Post Injection
Description: Lidocaine blood levels were obtained 30 minutes post injection micro g/L The difference between injection type- 95% confidence intervals for the difference between injection types was calculated. For the outcome variable, an assessment of treatment difference by subject, calculated as 1% Buffered minus 2% Non-Buffered, was performed using Wilcoxon rank sum tests with Proc NPAR1WAY (SAS v 9.3). Statistical significance was set as P < 0.05 for all outcomes.
Time Frame: 30 minutes post injection
Measure: Mean (Standard Deviation); unit: ug/L
Groups:
- Buffered Lidocaine and Non-Buffered Lidocaine: At Visit 1 each subject received Buffered Lidocaine anesthetic to block the inferior alveolar and lingual N; using Halstead or Gow-Gates techniques. No Buccal N. block. Venous blood samples were drawn from the antecubital fossa 30min post oral injection and assayed for blood lidocaine levels. Following a 2-week washout, subjects received Non-buffered Lidocaine in the same fashion at Visit 2.
Arm/Group | Buffered Lidocaine and Non-Buffered Lidocaine
Number analyzed (Participants) | 23
ug/L
  buffered lidocaine | 7.9 (16.2)
  non-buffered lidocaine | 15.8 (16.2)
Statistical Analysis 1: Comparison: Buffered Lidocaine and Non-Buffered Lidocaine; The difference between injection type- 95% confidence intervals for the difference between injection types was calculated. For the outcome variable, an assessment of treatment difference by subject, calculated as 1% Buffered minus 2% Non-Buffered, was performed using Wilcoxon signed rank tests (SAS v 9.3). Statistical significance was set as P < 0.05 for all outcomes; Test type: Other; p = 0.006, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -15, 95% CI 2-sided [-34.6 to -5.86] — for a cross over design difference in blood level was calculate buffered lidocaine minus non-buffered lidocaine

2. Secondary Outcome: Pain Intensity Scores
Description: Patients reported pain level immediately after injection of lidocaine via a Likert type scale where 1 = No Pain and 10 = Worst Pain Imaginable.
  For the outcome variable, an assessment of treatment difference by subject, calculated as 1% Buffered minus 2% Non-Buffered was performed.
Time Frame: Immediately after lidocaine injection
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buffered Lidocaine and Non-Buffered Lidocaine
Number analyzed (Participants) | 23
units on a scale
  buffered lidocaine | 2.6 (1.56)
  non-buffered lidocaine | 3.0 (2.2)
Statistical Analysis 1: Comparison: Buffered Lidocaine and Non-Buffered Lidocaine; The difference between injection type- 95% confidence intervals for the difference between injection types was calculated. For the outcome variable, an assessment of treatment difference by subject, calculated as 1% Buffered minus 2% Non-Buffered, was performed using ProcTTEST (SAS v 9.3). Statistical significance was set as P < 0.05 for all outcomes; Test type: Other; p = 0.096, t-test, 2 sided; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-1.46 to 0.13]

3. Secondary Outcome: Number of Minutes to Anesthesia Symptoms of Lower Lip
Description: Patients were instructed to record the time when they experienced the initial indication of anesthesia signs in the lower lip. This was reported as the number of minutes following nerve block injection.
  For the outcome variable, an assessment of treatment difference by subject, calculated as 1% Buffered minus 2% Non-Buffered was performed.
Time Frame: Patient report of anesthesia symptom onset following injection
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Buffered Lidocaine and Non-Buffered Lidocaine
Number analyzed (Participants) | 23
minutes
  buffered lidocaine | 10.2 (16.1)
  non-buffered lidocaine | 13.7 (16.1)
Statistical Analysis 1: Comparison: Buffered Lidocaine and Non-Buffered Lidocaine; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.23, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -1, 95% CI 2-sided [-4 to 1]

4. Secondary Outcome: Topical Anesthesia Effect Contralateral Lower Lip
Description: Investigator will administer 5-6 drops of the lidocaine to the contralateral lower lip and immediately ask if signs of numbness are present on the lip.
  Patients reported presence of numbness lower lip-Yes or No
Time Frame: At time of administration
Population: Unable to administer in this fashion because Lidocaine would not remain on lip surface therefore data were not collected
Arm/Group | Buffered Lidocaine and Non-Buffered Lidocaine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: two weeks
Groups:
- Buffered Lidicaine: In week One each subject would receive anesthetic to block the inferior alveolar and lingual N; Halstead or Gow-Gates techniques. No Buccal N. block.
  Venous blood samples would be drawn from the antecubital fossa 30min post oral injection and assayed for blood lidocaine levels
  Lidocaine: See above
- Non-bufered Lidocaine: In week One each subject would receive anesthetic to block the inferior alveolar and lingual N; Halstead or Gow-Gates techniques. No Buccal N. block. At least a week later injections would involve the alternate local anesthetic combination.
  Venous blood samples would be drawn from the antecubital fossa 30min post oral injection and assayed for blood lidocaine levels
  Lidocaine: See above
Arm/Group | Buffered Lidicaine | Non-bufered Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-30): https://cdn.clinicaltrials.gov/large-docs/83/NCT02620683/Prot_SAP_000.pdf